CLINICAL TRIAL: NCT05124210
Title: An Open-label, Non-comparator, Multicenter Study to Describe the Pharmacokinetics (PK), Pharmacodynamics (PD; Viral Load) and Safety Following a Single Intravenous or Intramuscular Dose of Sotrovimab in Pediatric Participants With Mild to Moderate COVID-19 at High Risk of Disease Progression
Brief Title: Pharmacokinetics, Pharmacodynamics, and Safety of Single-dose Sotrovimab in High-risk Pediatric Participants With Mild to Moderate COVID-19
Acronym: COMET-PACE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decrease in in-vitro neutralization of study drug against circulating SARS-CoV-2 variants
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215226
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; Pharmacokinetics; Safety; Pharmacodynamics; Sotrovimab; Pediatric; Intravenous; Intramuscular
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Sotrovimab Intravenous (IV) (6 to less than [<] 12 years) (Experimental): Participants in the age group 6 to < 12 years received up to a maximum of 500 milligram (mg) sotrovimab based on the body weight through Intravenous administration on Day 1
  Interventions: Biological: Sotrovimab
- Cohort A: Sotrovimab Intravenous (IV) (12 to less than [<] 18 years) (Experimental): Participants in the age group 12 to < 18 years received up to a maximum of 500 milligram (mg) sotrovimab based on the body weight through Intravenous administration on Day 1
  Interventions: Biological: Sotrovimab

INTERVENTIONS:
Biological: Sotrovimab — Sotrovimab will be administered.

SUMMARY:
This Phase 2b study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD) and safety of sotrovimab in pediatric participants from birth to less than (<)18 years old with mild-to-moderate Coronavirus Disease-2019 (COVID-19) at high risk of disease progression.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 32 weeks estimated gestational age (EGA), day of life (DOL) 0 to <18 years of age inclusive, at either the time of participant's signed assent (if age-appropriate) or parent(s)/legally authorized representative signing the informed consent.
* Participants with mild-moderate COVID-19.
* Participants at risk of disease progression with at least one of the following criteria: Age <1 year; Diabetes mellitus; Genetic or metabolic diseases; Obesity ); Cardiovascular disease; Sickle cell disease; Pulmonary disease; Neurologic disease; Immunosuppressed ; Baseline medical complexity (gastrostomy- or jejunostomy-dependence, parenteral nutrition dependence, tracheostomy-dependence, Baseline oxygen requirement, use of Continuous positive airway pressure [CPAP]/ Bilevel positive airway pressure [BiPAP]/ventilator support).

Exclusion Criteria

* Participant is pregnant or breastfeeding.
* Participant is currently hospitalized, or judged by the investigator as likely to require hospitalization in the next 24 hours, due to severe or critical COVID-19.
* Multisystem inflammatory syndrome in children (MIS-C).
* Prior, current, or planned future use of any of the following treatments during the study period: COVID-19 convalescent plasma, Monoclonal antibodies (mAbs) against Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) (for example [e.g.], casirivimab/imdevimab), intravenous immunoglobulin (IVIG) for any indication, or dexamethasone specifically for treatment of COVID-19.
* Current use of COVID-19 treatment (authorized, approved, or investigational).
* The following exclusions related to use of an authorized or approved vaccine for SARS-CoV-2 are applicable:

  1. Receipt of any authorized or approved vaccine for SARS-CoV-2 within 48 hours prior to dosing.
  2. Planned use of any authorized or approved vaccine for SARS-CoV-2 within 90 days of study drug administration per current Centers for Disease Control and Prevention (CDC) recommendations.
* Receipt of any non-SARS-CoV-2 vaccines within 14 days (for non-live vaccines) or 28 days (for live vaccine) of screening.
* Currently enrolled in another clinical study.
* Infants <24 weeks of age: maternal receipt of IVIG, SARS-CoV-2-directed convalescent plasma or SARS-CoV-2-directed mAb(s) within 3 months prior to birth or within 5 half-lives of the investigational product (whichever is longer).

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Cullman, Alabama
  - GSK Investigational Site, Mesa, Arizona

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 8 participants were enrolled in this study. Four age bands were planned to be enrolled (12 to less than 18 years, 6 to less than 12 years, 2 to less than 6 years and Birth to less than 2 years). Due to early termination of the study, no participants were enrolled in the 2 to less than 6 years and birth to less than 2 years age bands.
Pre-assignment Details: This study was conducted in 2 cohorts (Cohort A and Cohort B). The study was terminated, due to a decrease in in-vitro neutralization of sotrovimab against circulating Omicron BA.2 SARS-CoV-2 variants. Hence, Cohort B was not initiated. None of the participants received Intramuscular (IM) administration of sotrovimab.
Period: Overall Study
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Started | 3 | 5
Completed | 1 | 5
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years) | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 9.7 (0.58) | 14.2 (1.10) | 12.5 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 0 | 1 | 1
  WHITE | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Body Weight-Adjusted Serum Clearance (CL) of Sotrovimab
Description: Blood samples were collected at indicated timepoints and Pharmacokinetic (PK) analysis was performed. PK parameters were determined by population PK modelling method. The model considered the body weight of each participant to calculate the serum clearance of sotrovimab.
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: The analysis was performed on the PK Principal Stratum Set that included all participants in the PK analysis set who would be able to complete the IV dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per day (L/day)
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Liter per day (L/day) | 0.05 (27.6) | 0.10 (28.5)

2. Primary Outcome: Maximum Observed Concentration (Cmax) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods using Phoenix WinNonlin. The log-transformed data is transformed back to the original scale and presented here.
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: The analysis was performed on the PK Principal Stratum Set that included all participants in the PK analysis set who would be able to complete the IV dose. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 1 | 5
microgram per milliliter (µg/mL) | 342.96 (NA) — NA indicate that data is not available since only one participant was analyzed. Therefore Geometric Coefficient of Variation was not derived. | 191.67 (29.45)

3. Primary Outcome: Time to Reach Cmax (Tmax) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin.
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Day
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 1 | 5
Day | 0.000 [NA to NA] — NA indicate that data is not available since only one participant was analyzed, the full range (minimum and maximum) were not derived. | 0.003 [0.00 to 0.02]

4. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC[0-inf]) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated timepoints and Pharmacokinetic (PK) analysis was performed. PK parameters were determined by population PK modelling method.
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram per milliliter (day*ug/mL)
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Day*microgram per milliliter (day*ug/mL) | 6023.0 (7.91) | 4928.8 (24.4)

5. Primary Outcome: Terminal Elimination Half-Life (T1/2) Following Administration of Sotrovimab
Description: as for outcome 4
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Day | 37.5 (16.1) | 43.6 (22.0)

6. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) Following Administration of Sotrovimab
Description: Blood samples were collected at indicated timepoints and PK analysis was performed. PK parameters were determined by non-compartmental methods with Phoenix WinNonlin. The log-transformed data is transformed back to the original scale and presented here.
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 1 | 5
Liter | 1.42 (NA) — NA indicate that data is not available since only one participant was analyzed. Therefore Geometric Coefficient of Variation was not derived. | 5.49 (22.08)

7. Primary Outcome: Clearance (CL) Following Administration of Sotrovimab
Description: as for outcome 6
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per day (mL/day)
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 1 | 5
milliliter per day (mL/day) | 42.62 (NA) — NA indicate that data is not available since only one participant was analyzed. Therefore Geometric Coefficient of Variation was not derived. | 96.58 (30.44)

8. Primary Outcome: Relative Bioavailability (F) Following Administration of Sotrovimab
Description: as for outcome 3
Time Frame: Day 1 (End of Infusion), Day 5, 8 and 12, Week 12
Population: Due to early termination of the study, the Intramuscular (IM) administration cohort was not started. The bioavailability assessment was not performed between the Intravenous (IV) and Intramuscular (IM) administration of sotrovimab. Hence there is no data to report.
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. Protocol defined AESIs were included.
Time Frame: Up to Day 29
Population: The analysis was performed on the Safety Set (Cohort A) that included all participants who are exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Participants
  Participants with AE | 1 | 2
  Participants with SAE | 0 | 0
  Participants with AESI | 0 | 0

10. Secondary Outcome: Number of Participants With Progression of COVID-19 Through Day 29
Description: Progression of COVID-19 is defined as need for attended medical visit (including the visit to a hospital emergency room for management of illness or hospitalization for acute management of illness) or escalation to higher level of medical care or death.
Time Frame: Up to Day 29
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Development of Severe and/or Critical Respiratory COVID-19 Through Day 29
Description: Severe and/or critical respiratory COVID-19 as manifested by requirement for supplemental oxygen through Day 29. For participants who required oxygen or respiratory support for premorbid conditions, disease progression was defined as any sustained (greater than [>]24 hours) increase in the level or method of oxygen support required.
Time Frame: Up to Day 29
Population: The analysis was performed on the Virology Set (Cohort A) that included all participants who are exposed to study treatment and have a quantifiable SARS-CoV-2 viral load measurement at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

12. Secondary Outcome: Change From Baseline in Viral Load in Nasal Secretions Measured by Quantitative Reverse Transcriptase-Polymerase Chain Reaction (qRT-PCR)
Description: The viral load change from baseline in nasal secretions was measured by quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) at Day 5, Day 8, and Day 11.
Time Frame: Baseline (Day 1), at Day 5, Day 8 and Day 11
Population: The analysis was performed on the Safety Set (Cohort A) that included all participants who are exposed to study intervention. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 2 | 5
log10 copies per milliliter
  Baseline (Day 1) | 5.085 (0.2475) | 4.712 (1.0668)
  Day 5 | -1.270 (2.6304) | -2.160 (1.4053)
  Day 8 | -2.640 (0.6930) | -2.398 (1.6272)
  Day 11 | -3.305 (0.2475) | -2.870 (1.1430)

13. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI) Up to Week 36
Description: as for outcome 9
Time Frame: Up to Week 36
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
Number analyzed (Participants) | 3 | 5
Participants
  Participants with AE | 1 | 4
  Participants with SAE | 0 | 0
  Participants with AESI | 0 | 0

ADVERSE EVENTS:
Time Frame: Upto Week 36
Description: Safety Set comprised of all participants who are exposed to study treatment.
Arm/Group | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 1/3 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Sotrovimab Intravenous (IV) (6 to Less Than [<] 12 Years) (N=3) | Cohort A: Sotrovimab Intravenous (IV) (12 to Less Than [<] 18 Years) (N=5)
Hypoplastic left heart syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Polyomavirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05124210/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT05124210/SAP_001.pdf